CLINICAL TRIAL: NCT04414137
Title: Description of Eosinophilic Pneumonia in BJI/PJI Treated by Daptomycin
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 19-283
Record Dates: First submitted 2020-05-12; First posted 2020-06-04 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Dactinomycin Adverse Reaction; Bone and Joint Infection
Keywords: Eosinophilic pneumonia; Daptomycin; Bone and joint infection; Adverse event
MeSH Terms: conditions — Pulmonary Eosinophilia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Eosinophilic pneumonia on daptomycin: patients having an osteoarticular infection treated with daptomycin and which developped eosinophilic pneumonia
  Interventions: Other: Description of eosinophilic pneumonia due to daptomycine

INTERVENTIONS:
Other: Description of eosinophilic pneumonia due to daptomycine — Description of eosinophilic pneumonia in patients treated by daptomycin for an osteoarticular infection

SUMMARY:
Daptomycin is an antibiotic from the family of cyclic lipopeptides, bactericide, concentration-dependent. Its spectrum concerns Gram-positive bacteria.

Since the authorization of daptomycin in 2006, cases of eosinophilic pneumonia and pulmonary eosinophilia associated with its use have been reported in Europe and worldwide.

The purpose of this study is to describe the mechanism of occurrence of this AE with dapto; Prolonged exposure and accumulation at the alveolar level could potentially have a role. Better understanding the mechanisms of appearance of this AE would provide predictive elements making it possible to limit the occurrence of this AE in the future

DETAILED DESCRIPTION:
Daptomycin is an antibiotic from the family of cyclic lipopeptides, bactericide, concentration-dependent. Its spectrum concerns Gram-positive bacteria.

The Infectious Diseases Society of America recommends the use of daptomycin 6 mg / kg / day in the second-line treatment of IOA on staphylococcal but also enterococcal prostheses, as an alternative to vancomycin and linezolid.

In case of renal failure, daptomycin is often considered as a good therapeutic alternative to glycopeptides.

Since the authorization of daptomycin in 2006, cases of eosinophilic pneumonia and pulmonary eosinophilia associated with its use have been reported in Europe and worldwide. Although a large proportion of cases have been reported in patients receiving daptomycin in unapproved indications, the use of daptomycin in authorized indications has also been associated with this risk.

The dosage of daptomycin makes it possible to evaluate its effectiveness and prevent the occurrence of a overdose, provider of side effects.

The purpose of this study is to describe the mechanism of occurrence of this AE with dapto; Prolonged exposure and accumulation at the alveolar level could potentially have a role. Better understanding the mechanisms of appearance of this AE would provide predictive elements making it possible to limit the occurrence of this AE in the future

ELIGIBILITY:
Inclusion Criteria:

* patients having had an eosinophilic pneumonia under daptomycine given to treat an osteoarticular infection (BJI/PJI)

Exclusion Criteria:

-

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients having had an eosinophilic pneumonia under daptomycine given to treat an osteoarticular infection (BJI/PJI) treated at the CRIOAc Lyon
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-02-19 (Actual); Primary Completion 2021-01-20 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
description of BJI/BJI in patients having eosinophilic pneumonia due to daptomycin | 2 months
  description of the BJI/PJI (symptoms, type of evolution, type of implant)
description patients having eosinophilic pneumonia due to daptomycin | 2 months
  description of the patients (average age, medical background)
rate of eosinophilic pneumonia due to daptomycin in osteoarticular infection: the adverse event | 6 months
  number of cases and description of the adverse event as assessed by CTCAE v4.0
Evalutation of eosinophilic pneumonia due to daptomycin in osteoarticular infection: dosage of daptomycine | 6 months
  description of the use of daptomycine : dosage
Evalutation of eosinophilic pneumonia due to daptomycin in osteoarticular infection: duration of daptomycine | 6 months
  description of the use of daptomycine : duration
Evalutation of eosinophilic pneumonia due to daptomycin in osteoarticular infection: daptomycine plasma clearance | 6 months
  mean daptomycine plasma clearance (unit, liters per hour)
Evalutation of eosinophilic pneumonia due to daptomycin in osteoarticular infection: daptomycine volume distribution | 6 months
  mean daptomycine volume of distribution (unit, liters)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.crioac-lyon.fr/